CLINICAL TRIAL: NCT07176858
Title: EFFECT OF BRAIN GYM EXERCISES ON FUNCTIONAL ABILITIES IN CHILDREN WITH CEREBRAL PALSY
Brief Title: BRAIN GYM EXERCISES and CEREBRAL PALSY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Fahmy Hassan Al Nemr, assistant professor at faculty of physical therapy, Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004633
Record Dates: First submitted 2025-09-04; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy
Keywords: brain gym exercises; cognitive function; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- brain gym exercises and designed physical therapy program (Experimental)
  Interventions: Other: brain gym exercise
- designed physical therapy program (Experimental)
  Interventions: Other: specially designed pt program

INTERVENTIONS:
Other: brain gym exercise — specially designed physical therapy program in addition to brain gym exercises for 60 min (30 min designed P.T program and other 30 min for brain gym exercises), 3 sessions/ week for 3 successive months. eight Brain Gym exercises will be selected: Cross Crawl, Lazy 8s, Hook-ups, Brain Buttons, The Elephant, The Owl, Neck Rolls, Double Doodle
  Arms: brain gym exercises and designed physical therapy program
Other: specially designed pt program — conventional physical therapy program including reinforcement of the normal motor development, reflex inhibiting patterns, postural reaction, stretching, strengthening exercises, and gait training was applied to children in the control group
  Arms: designed physical therapy program

SUMMARY:
Brain gym is a series of exercises developed to enhance learning by improving cognitive function and fostering a stronger mind-body connection. It uses physical and mental techniques to stimulate both hemispheres of the brain. This approach is rooted in kinesiology and applied neuroscience, fields that study the relationship between bodily movements and brain activity.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of spastic hemiplegic CP
2. Degree of spasticity ranges from 1 and 1+, according to modified Ashworth scale (MAS)
3. The age of the selected children will range from 6 to 8 years old.
4. Children are levels I and II according to GMFCS

Exclusion Criteria:

1 - Children with visual or auditory problems. 2. Children with severe intellectual disability (IQ less than 65 according to Stanford Binet intelligence scale).

3. Children have been injected with Botox injection or have done surgery in the last 6 months

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-10-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
cognitive functions will be measured by computer-based RehaCom software. It is a valid and reliable tool. higher score indicate worse results | 3 month
The quality of life of all children will be assessed by pediatric quality of life scale which is a valid and reliable scale to assess quality of life in CP children. higher scores indicate better results. raw scores range from 0 to 100 | 3 month

IPD SHARING:
Plan to Share IPD: No